CLINICAL TRIAL: NCT06487923
Title: The Effects of Knowledge and Awareness of Pelvic Floor Health on Dyspareunia in Postpartum Women
Brief Title: Knowledge and Awareness of Pelvic Floor Health
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Other Study IDs: E-22686390-050.99-34849
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Floor Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum Women: 298 primiparous women who have given birth vaginally in the last year

SUMMARY:
The aim of this study is to investigate the relationship between knowledge and awareness of pelvic floor health and dyspareunia, pelvic floor dysfunctions, and quality of life in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Being a native speaker of Turkish
* Being in the first year of postpartum
* Women who had a vaginal delivery
* Primiparous women
* Women aged 18 and over

Exclusion Criteria:

* Women who have not given birth
* Multiparous women
* Women who had a cesarean delivery
* Having difficulty to understanding evaluations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Primiparous women who have given birth within the past year aged 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Health Knowledge Quiz | Baseline
  This scale is a self-report tool developed to measure pelvic floor knowledge and awareness.The scale was developed by Wala'a Al-Deges in 2019. The original version is in Turkish. It consists of 29 questions divided into 3 sub-parameters. A high score indicates a high level of awareness.
Carol Postpartum Sexual Function And Dyspareunia Assessment Scale | Baseline
  This scale is a self-report tool developed to evaluate sexual functions and dyspareunia who have resumed vaginal intercourse after vaginal delivery. It developed by Pérez-García, Solís-Muñoz. Turkish Validity and reliability study was conducted by Evili. The scale consists of 11 items and 4 subparameters in a Likert-type format. Except for 'preparation for sexual activity', a high score indicates a high level of dysfunction.
Sociodemographic Information Form | Baseline
  The demographic information form consisted of 27 questions to determine and classify individuals' socio-demographic characteristics, including descriptive features such as age, height, weight, BMI, marital status, recorded using this form.

SECONDARY OUTCOMES:
Nottingham Health Profile | Baseline
  This scale assesses individuals' well-being in physical, emotional, and social domains. It Developed by Hunt in 1981. Turkish Validity and reliability study was conducted by Kucukdeveci in 2000. The scale consists of 38 items and 6 subparameters. A high score indicates a low quality of life.
Prolapse and Incontinence Knowledge Questionnaire | Baseline
  To assess individuals' knowledge levels about prolapse and incontinence, the Prolapse and Incontinence Knowledge Questionnaire was used. Validity and reliability studies of the questionnaire were conducted by Celenay in 2019. The questionnaire consists of a total of 24 statements, with 12 statements related to Pelvic Organ Prolapse and 12 statements related to Urinary Incontinence. Correct responses contribute to the total score, which ranges from a minimum of 0 to a maximum of 12. A higher score indicates greater knowledge about incontinence and prolapse.
Global Pelvic Floor Symptom Bother Questionnaire | Baseline
  The Global Pelvic Floor Dysfunction Inventory is used to assess whether individuals have any pelvic floor dysfunctions such as urinary urgency and frequency, difficulty emptying the bladder, pelvic organ prolapse, difficulty with defecation, fecal incontinence, sexual dysfunction, and to evaluate the degree of discomfort caused by these conditions if present. Validity and reliability study in Turkish women was conducted by Dogan in 2015. It consists of 9 questions. The total score from the questionnaire ranges from 0 to 45, with a higher score indicating a higher degree of discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)